CLINICAL TRIAL: NCT03494348
Title: Aspects of Alignment, Function, and Migration Behaviour in Two Conceptually Different Articular Surface Designs in the Cruciate Retaining Version of the Cemented Persona Knee System - A Randomized Study Evaluated by RSA and CT Analysis
Brief Title: RSA Study of Persona TKA With CR vs MC Polyethylene
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Region Skane (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Persona RSA study_MT
Record Dates: First submitted 2018-04-03; First posted 2018-04-11 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Radiostereometry (RSA); Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cruciate Retaining Polyethylene (CR) (No Intervention): This is the standard Polyethylene articular surface
- Medial Congruent Polyethylene (MC) (Active Comparator): The intervention here will be the MC articular surface. This is the new Polyethylene articular surface with a more congruent medial side and a more flat lateral side which should better resemble natural anatomy.
  Interventions: Device: Medial Congruent Polyethylene (MC)

INTERVENTIONS:
Device: Medial Congruent Polyethylene (MC) — One group receives the conventional CR surface and the other the new MC articular surface
  Other Names: MC
  Arms: Medial Congruent Polyethylene (MC)

SUMMARY:
The aim of this study is to evaluate, over a 2 year period, the migration pattern, function and the possibility of anatomical reconstruction of a relatively new total knee arthroplasty (TKA) concept, the Persona. Sixty patients will be randomized into 2 groups of 30 patients each, with one group receiving the Persona TKA with a conventional Cruciate Retaining (CR) polyethylene articular surface and the other group with a newly developed Medial Congruent (MC) articular surface. Patients will be followed up with Radiostereometry (RSA), conventional radiography, outcome questionnaires, clinical evaluation and Computer Tomography (CT). The migration pattern of the components will be evaluated as well as the degree of anatomical reconstruction and clinical result.

We plan also to do a 5 year follow-up of the patients with RSA and PROMS.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee necessitating knee replacement
* ASA I-III
* BMI 18 - 35

Exclusion Criteria:

* Joint sepsis in history
* immunosuppresive drugs last 5 years
* Rheumatoid arthritis
* Severe osteoporosis or other metabolic bone diseases
* Neuromuscular diseases
* Personal disorders suspected of limiting rehab and completion of the trial period
* Previous osteotomy of affected limb
* Intra-articular knee fracture of affected limb
* Peroperative fracture
* Severe deformity of affected joint in need of augmentation or excessive release
* Obvious need for more constrained knee than CR

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Radiostereometry (RSA) | First postoperative day, 3 months, 1 year, 2 years and 5 years
  Measure the change in component migration over time (translation and rotation around the x-, y- and z-axis)

SECONDARY OUTCOMES:
Computer Tomography (CT) | Preoperatively and 3 months postoperatively
  Measure the preoperative malalignment of the knee and the postoperatively achieved alignment and achieved prosthesis position
Conventional radiography | Preoperatively and 3 months postoperatively
  Measure the preoperative malalignment of the knee and the postoperatively achieved alignment and achieved prosthesis position
General health questionnaire | Preoperatively, 1, 2 and 5 years postoperatively
  EuroQol (EQ-5D) -standardized instrument for use of general health outcome
Knee specific health questionnaire | Preoperatively, 1, 2 and 5 years postoperatively
  Knee disability and Osteoarthritis Outcome Score (KOOS) - this is a knee specific questionnaire measuring patients knee function and pain situation

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Flivik, MD PhD, Principal Investigator — Dept of Orthopedics, Skåne University Hospital
Locations (1):
- Department of Orthopedics, Skane University Hospital, Lund University, Lund, Sweden